CLINICAL TRIAL: NCT00237757
Title: Rehabilitation Team Functioning and Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: O3225-R
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Stroke
Keywords: Patient Care Team; Rehabilitation outcomes; Treatment outcomes
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): The experimental arm consisted of a six month staff training period with an emphasis on effective team functioning to improve patient outcomes. The core of the intervention consisted of a concentrated 2.5 day workshop in Atlanta for 29 rehabilitation team leaders from 15 VA hospitals. Several weeks after the workshop, participants received a custom action plan developed on issues discussed in the workshop. The experimental arm also received a summary of results of the initial survey along with comparative data from all other sites. During the subsequent 5 months after the workshop, research staff maintained regular contact with research participants through telephone and videoconferencing
  Interventions: Behavioral: Information feedback
- Arm 2 (Active Comparator): The comparison arm (staff on 16 teams) completed the identical summary of staff, hospital, and team characteristics. The local PIs at the Comparison sites received summaries of the survey findings, comparative data from other participating VA sites, and suggestions on how this information could be used to improve patient outcomes. In addition, participants in the comparison arm were invited to contact the research staff for help in interpreting data or to set-up a process improvement initiative.
  Interventions: Behavioral: Information feedback

INTERVENTIONS:
Behavioral: Information feedback — The experimental arm consisted of a six month staff training period. The core of the intervention consisted of a concentrated 2.5 day workshop in Atlanta for 29 rehabilitation team leaders from 15 VA hospitals. Several weeks after the workshop, participants received a custom action plan developed on issues discussed in the workshop. The experimental arm also received a summary of results of the initial survey along with comparative data from all other sites. During the subsequent 5 months after the workshop, research staff maintained regular contact with research participants through telephone and videoconferencing. The comparison arm (staff on 16 teams) completed the identical summary of staff, hospital, and team characteristics. The local PIs at the Comparison sites received summaries of the survey findings, comparative data from other participating VA sites, and suggestions on how this information could be used to improve patient outcomes.
  Arms: Arm 1
Behavioral: Information feedback — The comparison arm (staff on 16 teams) completed the identical summary of staff, hospital, and team characteristics. The local PIs at the Comparison sites received summaries of the survey findings, comparative data from other participating VA sites, and suggestions on how this information could be used to improve patient outcomes. In addition, participants in the comparison arm were invited to contact the research staff for help in interpreting data or to set-up a process improvement initiative.
  Arms: Arm 2

SUMMARY:
The purpose of the study is to determine if 1. Rehabilitation staff can be trained to work better together as a team; and 2. Better team work improves patient outcomes.

DETAILED DESCRIPTION:
The benefits of team treatment are widely accepted. Prior research has shown that how rehabilitation teams go about their work makes a difference in the patients they treat. However, there is little information about what, specifically, the team does that results in patients who are able to do more for themselves. The objectives of this clinical trial was to test whether a team training intervention in stroke rehabilitation was associated with improved patient outcomes. We conducted a cluster randomized trial of 31 rehabilitation units comparing stroke outcomes between intervention and control groups. in thirty-one VA medical centers with 237 clinical staff on 16 control teams and 227 staff on 15 intervention teams. There were 487 stroke patients treated by these teams before and after the intervention.

The intervention consisted of a multiphase, staff training program delivered over six months, including: an off-site workshop emphasizing team dynamics, problem solving, and the use of performance feedback data; and action plans for process improvement; and telephone and videoconference consultations. Control and intervention teams received site- specific team performance profiles with recommendations to use this information to modify team process.

The main outcomes measures consisted of three patient outcomes: functional improvement as measured by the change in motor items of Function Independence Measure (FIM), community discharge, and length of stay (LOS). For both the primary (stroke only) and secondary analyses (all patients), there was a significant difference in improvement of functional outcome between the two groups, with the percentage of stroke patients gaining more than a median FIM gain of 23 points increasing significantly more in the intervention group (difference in increase = 13.6%, P=0.032). There was no significant difference on LOS or rates of community discharge. Stroke patients treated by staff who participated in a team training program were more likely to make functional gains than those treated by staff receiving information only. This study is a randomized cluster trial which tested used workshops to train rehabilitation staff. Patients treated by trained teams were compared with patients treated by teams that did not have workshop training. Stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Randomized, controlled subjects were VA inpatient rehabilitation teams. Secondary data included telephone surveys from discharged patients treated by the rehabilitation teams.

Exclusion Criteria:

* VA sites which did not submit data to the VA-FSOD - the national functional outcomes database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
functional gain as measured by motor FIM score | One year post team training intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dale Christian Strasser, MD, Principal Investigator — VA Medical Center, Decatur
Locations (1):
- VA Medical Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- [Background] Strasser DC, Falconer JA, Uomoto JM. Can quality of care indicators measure quality of care? Arch Phys Med Rehabil. 2012 Nov;93(11):2130-1; author reply 2131-2. doi: 10.1016/j.apmr.2012.04.035. No abstract available. PMID 23101971
- [Background] Stevens AB, Strasser DC, Uomoto J, Bowen SE, Falconer JA. Utility of Treatment Implementation methods in clinical trial with rehabilitation teams. J Rehabil Res Dev. 2007;44(4):537-46. doi: 10.1682/jrrd.2006.09.0120. PMID 18247250
- [Background] Strasser DC, Uomoto JM, Smits SJ. The interdisciplinary team and polytrauma rehabilitation: prescription for partnership. Arch Phys Med Rehabil. 2008 Jan;89(1):179-81. doi: 10.1016/j.apmr.2007.06.774. PMID 18164351
- [Background] Strasser DC, Smits SJ, Falconer JA, Herrin JS, Bowen SE. The influence of hospital culture on rehabilitation team functioning in VA hospitals. J Rehabil Res Dev. 2002 Jan-Feb;39(1):115-25. PMID 11926323
- [Result] Strasser DC, Falconer JA, Herrin JS, Bowen SE, Stevens AB, Uomoto J. Team functioning and patient outcomes in stroke rehabilitation. Arch Phys Med Rehabil. 2005 Mar;86(3):403-9. doi: 10.1016/j.apmr.2004.04.046. PMID 15759219
- [Result] Strasser DC, Burridge AB, Falconer JA, Herrin J, Uomoto J. Measuring team process for quality improvement. Top Stroke Rehabil. 2010 Jul-Aug;17(4):282-93. doi: 10.1310/tsr1704-282. PMID 20826416
- [Result] Strasser DC, Falconer JA, Stevens AB, Uomoto JM, Herrin J, Bowen SE, Burridge AB. Team training and stroke rehabilitation outcomes: a cluster randomized trial. Arch Phys Med Rehabil. 2008 Jan;89(1):10-5. doi: 10.1016/j.apmr.2007.08.127. PMID 18164324
- [Result] Smits SJ, Falconer JA, Herrin J, Bowen SE, Strasser DC. Patient-focused rehabilitation team cohesiveness in veterans administration hospitals. Arch Phys Med Rehabil. 2003 Sep;84(9):1332-8. doi: 10.1016/s0003-9993(03)00197-7. PMID 13680570
- [Derived] Strasser DC, Burridge AB, Falconer JA, Uomoto JM, Herrin J. Toward spanning the quality chasm: an examination of team functioning measures. Arch Phys Med Rehabil. 2014 Nov;95(11):2220-3. doi: 10.1016/j.apmr.2014.06.013. Epub 2014 Jul 4. PMID 25007707